CLINICAL TRIAL: NCT05813899
Title: Efficacy of Lactobacillus Paracasei PS23 for Patients With Post-COVID-19 Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The covid-19 epidemic was calming down and not many people were suffering from the post covid 19 syndrome
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 22CT054be
Record Dates: First submitted 2023-04-11; First posted 2023-04-14 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Post-COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat-treated PS23 (Experimental): PS23 heat-treated, 2 caps daily use
  Interventions: Dietary Supplement: PS23 heat-treated
- Placebo (Placebo Comparator): The placebo , 2 caps daily use
  Interventions: Dietary Supplement: PS23 heat-treated

INTERVENTIONS:
Dietary Supplement: PS23 heat-treated — PS23 heat-treated, 2 caps daily use

SUMMARY:
To evaluate whether probiotics PS23 can improve the symptoms of patients with long COVID-19 ; also to evaluate the effects on blood cortisol and inflammation-related indicators in patients.

DETAILED DESCRIPTION:
It is expected that a total of 120 subjects will be recruited within 3 years after IRB approval, divided into two groups of 60 subjects, respectively consuming PS23 heat-treated bacteria or placebo, and completing the 6-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged above 20 years old and below 65 years old.
2. Those who consciously have long COVID-19 symptoms or actively respond to website advertisements to express interest in participating in this clinical researcher.
3. Those who received the confirmation SMS or the COVID-19 rapid test positive 4 weeks ago.

Exclusion Criteria:

1. Have taken antibiotics within one month or are receiving antibiotic treatment.
2. Have taken probiotic products have been used within two weeks (excluding yogurt, yogurt, Yakult and other related foods).
3. Cancer or immunocompromised patients undergoing treatment.
4. Those who are allergic to lactic acid bacteria products.
5. Diagnosed with dementia before being diagnosed with COVID-19.
6. Prior to or currently taking medication for acute or psychiatric illness prior to the diagnosis of COVID-19.
7. The investigator judges that it is not suitable to participate in the researcher.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression scales of Severity rated by clinician（CGI） | From Baseline to 6 Weeks Assessed
  The CGIC is a single-item questionnaire that asks the investigator to assess a patient's TD symptoms at specific visits after initiating therapy. The CGIC uses a 7 point Likert Scale, ranging from very much worse (-3) to very much improved (+3), to assess overall response to therapy. A treatment success was defined as "much improved" or "very much improved" at the week 6 visit.

SECONDARY OUTCOMES:
Wechsler Adult Intelligence Scale 4th version | From Baseline to 6 Weeks Assessed
  The WAIS-IV is a measure of cognitive function in older adolescents and adults. Participants complete the Digit Span subtest, which measures auditory working memory for numerical information.
Color Trails Test（CTT） | From Baseline to 6 Weeks Assessed
  There are two subtests: CTT1 & CTT2. The time spend to complete the two subtest is used representing executive function of the participants.
Insomnia Severity Index（ISI） | From Baseline to 6 Weeks Assessed
  The Insomnia Severity Index (ISI) is a brief instrument that was designed to assess the severity of both nighttime and daytime components of insomnia.
The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16, QLESQ-16 | From Baseline to 6 Weeks Assessed
  The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16 (QLESQ-16) is a valid, reliable self-report instrument for assessing quality of life.
State and Trait Anxiety Index (STAI) | From Baseline to 6 Weeks Assessed
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Patient Heath Questionnaire-9 (PHQ-9) | From Baseline to 6 Weeks Assessed
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression: The PHQ-9 incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool.Depression Severity: 0- none, 1-4 minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. Validity has been assessed against an independent structured mental health professional (MHP) interview. PHQ-9 score ≥10 had a sensitivity of 88% and a specificity of 88% for major depression.
Visual Analogue Scale-GI (VAS-GI) | From Baseline to 6 Weeks Assessed
  Visual Analogue Scale for GI symptoms, VAS-GI (visual analogue scale, VAS 0-10) was designed to measure the response of symptoms and well-being in patients after taking probiotics or placebo.
Patient Global Impression scales of Improvement rated by patient（PGI-C） | From Baseline to 6 Weeks Assessed
  The PGIC consists of one item taken from the clinical global impression and adapted to the patient. The minimum total score possible is 1 and the maximum total score possible is 7. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided